CLINICAL TRIAL: NCT01742442
Title: Cancer in the Elderly: Prevalence and Impact of Age Related Problems. A Prospective Observational Study
Brief Title: Cancer in the Elderly: Prevalence and Impact of Age Related Problems
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Oslo University Hospital (Other); Diakonhjemmet Hospital (Other); Vestre Viken Hospital Trust (Other); University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: E12224; 2012/104 C (Other: Regional Ethical Review Board HSO, Norway)
Record Dates: First submitted 2012-11-26; First posted 2012-12-05 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2017-09

CONDITIONS: Cancer
Keywords: Cancer; elderly OR older; chemotherapy; geriatric assessment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (serum and EDTA blood) for analysis of inflammatory markers. Dependent on the study results and results from other studies that may emerge during the study conduct, analyses of other markers of ageing may also be conducted
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older cancer patients: Older cancer patients 70 years or older referred to specialist oncology outpatient clinics

SUMMARY:
About 50% of cancer patients are >70 years at diagnosis. Age related somatic and psychiatric problems may influence the course of cancer and its treatment. The present study is a prospective observational study. Age related problems will be assessed by clinical frailty indicators covering areas that are recommended in geriatric oncology. The aim is to describe the frequency of age related problems in a cohort of Norwegian cancer patients > 70 years of age, to investigate the predictive/prognostic impact of these indicators on cancer and treatment related morbidity and mortality, and to investigate the association between clinical frailty indicators, sarcopenia (severe loss of muscle mass) and inflammatory response. Patients are recruited at outpatient cancer services, Innlandet Hospital HF (SI), Oslo University Hospital, and Akershus University Hospital. Estimated sample size is 300 with 30 months inclusion and 2 years follow-up. The study emerges from SI in collaboration with several external national and international centres

DETAILED DESCRIPTION:
The proportion of elderly cancer patients is high and is likely to increase due to an increasing cancer incidence and an aging population. The prevalence and impact of age related problems are, however, poorly documented, and elderly patients may therefore be subjects to under-treatment and arbitrary modifications of treatment regimens. In order to improve clinical practice, precise identification of patients with increased vulnerability and risk of adverse outcomes is paramount.

In the present study, eligible patients will be identified by referral to oncology services at one of the participating cancer units. After consent, the baseline registrations will be performed including relevant medical and sociodemographic data, and quality of life. Age related problems will be assessed by clinical indicators covering comorbidity, medication, emotional, physical and cognitive function and nutritional status. Muscle mass will be quantified by analyses of diagnostic CT scans and a biobank will be established for the analyses of inflammatory markers. Upon inclusion, the patients' physician will be asked to rate the patients as fit, frail or intermediate according to the physicians' subjective judgement. The patients will be followed with assessments of quality of life, emotional function and nutritional status (self-report), cognitive and physical function (self-report and performance tests), muscle mass (diagnostic CT scans when available) and inflammatory markers (biobank). Follow up data will also include registry data (hospital records, primary health care registries, The Norwegian Patient Registry, The Norwegian Cancer Registry and the Norwegian Cause of Death registry). We will describe the prevalence of age related problems, investigate the relation between clinical frailty indicators, sarcopenia, inflammatory response and the physicians' subjective evaluation of the patients' health status. The predictive/prognostic impact of frailty indicators on the patients' self-reported physical function and quality of life, hospital and nursing home admittance, treatment toxicity and survival will also be investigated

ELIGIBILITY:
Inclusion Criteria:

* age >= 70 years
* histologically/cytologically verified cancer disease
* referred to specialist oncology service
* no former chemotherapy for actual status (new cancer diagnosis no former or chemotherapy for metastatic disease)
* subject to medical oncological treatment that may be initiated and administered at the hospital trust the patient is referred to
* able to provide written consent
* fluent in Norwegian (orally and written)

Exclusion Criteria:

- lymphomas and haematological malignancies

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Consequetive patients referred to a specialist outpatient clinic for medical cancer treatment
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of age related problems | At baseline
  Age related problems assessed by clinical indicators including comorbidity, medication, emotional, physical, cognitive function, nutritional status and quality of life
Physical decline | Follow-up
  Physical decline during follow-up, as measured by the EORTC QLQ-C30 questionnaire. We will investigate the predictive value of frailty (measured by clinical indicators), sarcopenia and inflammatory response on this outcome. Primary endpoint is defined as 2 months of follow-up

SECONDARY OUTCOMES:
Hospital and nursing home admittance | 2-4 months and 2 years follow-up
  The predictive value of frailty indicators (including clinical indicators, sarcopenia and inflammatory response) on the outcome
Quality of life | 2 - 4 months and 2 years follow-up
  The predictive impact of frailty indicators (including clinical indicators, sarcopenia and inflammatory response) on the outcome
Treatment toxicity | 2-4months and up to 2 years
  The predictive impact of frailty indicators (including clinical indicators, sarcopenia and inflammatory response) on the outcome "treatment toxicity" defined in terms of any adverse event requiring hospital admission and haematological toxicity (grade 3-4 cytopenia). Toxicity during the first course of chemotherapy (2-3 weeks), during 3-4 courses (2-3 months) and for the whole follow-up. i.e. up to 2 years will be investigated
survival | 2 years follow-up
  The prognostic value of frailty indicators (including clinical indicators, sarcopenia and inflammatory response on the outcome

OTHER OUTCOMES:
The association between clinical frailty indicators, sarcopenia and inflammatory response | Baseline and 2 years follow-up
  Association between clinical frailty indicators, sarcopenia and inflammatory response
The association between physicians' subjective evaluation of the patients' health status and clinical frailty indicators | Baseline and 2 years follow-up
  Agreement between physicians evaluation of health status and frailty based on a systematic assessment of frailty indicators

CONTACTS AND LOCATIONS:
Overall Officials: Marit S Jordhøy, MD, PhD, Principal Investigator — Sykehuset Innlandet and Oslo University Hospital; Siri Kristjansson, MD, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (3):
- Norway (3):
  - Akershus University Hospital, Lillestrøm, Lørenskog
  - Innlandet Hospital Trust, Brumunddal
  - Oslo University Hospital Ullevål, Oslo

REFERENCES:
- [Background] Hurria A, Togawa K, Mohile SG, Owusu C, Klepin HD, Gross CP, Lichtman SM, Gajra A, Bhatia S, Katheria V, Klapper S, Hansen K, Ramani R, Lachs M, Wong FL, Tew WP. Predicting chemotherapy toxicity in older adults with cancer: a prospective multicenter study. J Clin Oncol. 2011 Sep 1;29(25):3457-65. doi: 10.1200/JCO.2011.34.7625. Epub 2011 Aug 1. PMID 21810685
- [Background] Kristjansson SR, Nesbakken A, Jordhoy MS, Skovlund E, Audisio RA, Johannessen HO, Bakka A, Wyller TB. Comprehensive geriatric assessment can predict complications in elderly patients after elective surgery for colorectal cancer: a prospective observational cohort study. Crit Rev Oncol Hematol. 2010 Dec;76(3):208-17. doi: 10.1016/j.critrevonc.2009.11.002. Epub 2009 Dec 14. PMID 20005123
- [Derived] Kirkhus L, Harneshaug M, Saltyte Benth J, Gronberg BH, Rostoft S, Bergh S, Hjermstad MJ, Selbaek G, Wyller TB, Kirkevold O, Borza T, Saltvedt I, Jordhoy MS. Modifiable factors affecting older patients' quality of life and physical function during cancer treatment. J Geriatr Oncol. 2019 Nov;10(6):904-912. doi: 10.1016/j.jgo.2019.08.001. Epub 2019 Aug 21. PMID 31444088